CLINICAL TRIAL: NCT05262465
Title: A Multicenter Clinical Study of Microtransplantation Combined With Azacytidine to Improve the Efficacy of Elderly Acute Myeloid Leukemia
Brief Title: Microtransplantation Combined With Azacytidine to Improve the Efficacy of EAML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: guomei (Other)
Responsible Party: Sponsor-Investigator, guomei, director, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Organization: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MST-EAML2020
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MST for unfit (Experimental): Induction chemotherapy can use azacytidine combined with low-dose cytarabine, or azacytidine combined with BCL / 2 inhibitor, and infuse modified peripheral blood hematopoietic stem cells after chemotherapy.
  Consolidation chemotherapy used azacytidine combined with low-dose cytarabine. After chemotherapy, modified peripheral blood hematopoietic stem cells were infused and repeated for 3 courses.
  Interventions: Biological: microtransplantation, HLA-mismatched donor peripheral stem cell infusion; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Biological: microtransplantation, HLA-mismatched donor peripheral stem cell infusion — HLA-mismatched donor peripheral stem cell infusion
  Other Names: DSI
Drug: Azacitidine — azacytidine 50-75mg/m2
  Other Names: Demethylated drugs
Drug: Venetoclax — Venetoclax 100-300mg/d ×3d，400mg 4-28d
  Other Names: BCL/2 inhibitor

SUMMARY:
Patients enrolled from each center according to confirmed criteria specified in cooperative scheme are recieved induction and consolidation chemotherapy with microtransplantation . Observe the remission rate and 2-year disease-free survival (DFS) and overall survival(OS) rate.

DETAILED DESCRIPTION:
Microtransplantation, which combines chemotherapy with adoptive infusion of granulocyte colony stimulating factor (G-CSF) mobilized HLA-mismatched peripheral blood stem cells (GPBSC). Data from more than 70 elderly AML patients who received microtransplantation in Beijing showed that the remission rate and 2-year disease-free survival (DFS) reach 75-82% and 32-39% respectively, and microchimerisms (donor cells<1%) were detected without GVHD. The results have been clinically validated in several other centers in China, United States and Australia.

In this study, azacytidine, decitabine, BCL / 2 inhibitor and other drugs combined with micro transplantation were used in elderly AML in order to improve the curative effect.

Patients enrolled from each center according to confirmed criteria specified in cooperative scheme are recieved induction and consolidation chemotherapy with microtransplantation . Observe the remission rate and 2-year disease-free survival (DFS) and overall survival(OS) rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have elderly (60-85 ages) AML pathologically confirmed per WHO guidelines.
* Patients have not been treated before.
* Patients must have ECOG Performance status of 0,1,or 2. If ECOG 2.
* Patients must have a HLA mismatched donor who should be able to provide informed consent.
* All genders and races are eligible.
* ALT and AST≤3 ×ULN, TBIL≤1.5 × ULN, Cr≤2 ×ULN or CrCl≥40 mL/min
* By means of ultrasonic Heartbeat map or multiple gated acquisition (MUGA) scanning determination of LVEF in the normal range.
* Donors must be able to safely undergo leukapheresis.

Exclusion Criteria:

* received operation 4 weeks before randomization
* acute promyelocytic leukemia,Myeloid sarcoma, chronic myeloid leukemia in accelerated phase and blastic phase;
* active CNS disease, pregnancy, or other major medical or psychiatric illnesses that could compromise tolerance to this protocol
* occurred stroke or intracranial hemorrhage within 6 months before randomization.
* Require the use of warfarin or equivalent of vitamin K antagonists (such as phenprocoumon) anticoagulant.
* There is clinical significance of cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months before randomization, or any heart function grade 3 (moderate) or 4 (severe ) heart disease in accordance with the functional classification method of New York Heart Association (NYHA).
* Known to have the following history: human immunodeficiency virus (HIV) or active hepatitis C virus or hepatitis B virus infection
* Any situation processed by the PI that will be damaged to the patients safety.
* Patients and / or authorized family member refuse to sign the consent.
* attend other clinical researchers in 3 months.
* Donors exclusion criteria include:active infection or malignancy, cardiovascular instability, severe anemia, severe coagulation disorder, pregnancy, inadequate venous access, inability to provide consent, or any other condition deemed unsafe by the treatment staff.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
the remission rate | 2month
  ①bone marrow: blasts <5% (with a count of at least 200 Nucleated cells).②Hemogram: absolute neutrophil count of more than 1.0×109/L，platelets of >100×109/L. ③Clinical: Without the signs and symptoms caused by leukemia infiltration d , and independent of transfusion;

SECONDARY OUTCOMES:
Disease Free Survival | 2 year
  Measured from complete remission to the date of death or the date of last follow-up examination;
Overall Survival | 2 year
  measured from the Date of beginning therapy to the date of death or the date of last follow-up examination;

OTHER OUTCOMES:
treatment-related mortality | 2 year
  Early mortality: death within 4 weeks after initiation of induction therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The fifth medical center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No